CLINICAL TRIAL: NCT04747067
Title: The Effect of Hemodiafiltration Versus High Flux Dialysis On Free Light Chains Reduction And Its Relation To Albumin Loss.
Brief Title: To Assess the Effect of HDF Versus High Flux Dialysis on Free Light Chains and Cumulative Albumin Loss, in End Stage Renal Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Reem Sultan, Assistant lecturer of Internal Medicine and Nephrology, Ain Shams University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HD vs HDF
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: End Stage Renal Disease; Hemodiafiltration; Hemodialysis
Keywords: End stage renal disease (ESRD); hemodiafiltration (HDF); hemodialysis (HD); Free light chains; Albumin loss; Kappa and lambda
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: It is a pilot crossover study, 25 ESRD patients were dialyzed using dialyzer; BIOPURE 260 HF on a single session on two hemodialysis modalities (conventional HD and online post-dilution HDF) with washout period of 2 weeks using high flux dialyzers with maximum surface area 2.0 m2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-flux Hemodialysis (Experimental): patients treated by conventional hemodialysis
  Interventions: Device: BIOPURE 260HF dialyzer
- Hemodiafiltration (Experimental): patients treated by online post-dilution hemodialysis
  Interventions: Device: BIOPURE 260HF dialyzer

INTERVENTIONS:
Device: BIOPURE 260HF dialyzer — Dialyzer with effective surface area 2.6 m2, High-flux polyethersulfone hollow fiber with steam sterilization, myoglobin sieving coefficient (SC) 0.7, membrane cutoff 40,000 Daltons (Allmed Medical Gmbh)

SUMMARY:
Removal of uremic toxins is the main goal of HD, It was improved by using high volume convective technique with high flux (HF) dialyzer. This technique removes medium - large molecular weight solutes giving higher dialysis adequacy and consequently improving the quality of life.

This study will assess the effect of hemodiafiltration (HDF) versus high flux dialysis on free light chains (FLC) reduction as a marker of HD adequacy and its relation to albumin loss using dialyzer effective surface area 2.6m2.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent HD patients on regular hemodialysis sessions for >6 months 3 sessions/week of 4 hours duration.
* Patients with Arterio-venous fistula as dialysis access.

Exclusion Criteria:

* Patients with hemodialysis catheters.
* Patients with active inflammation or infection.
* Decompensated heart failure.
* Liver Cell Failure ( Child B,C)
* Patients with known malignancies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Free light chain reduction | 1 day of hemodialysis session
  Measurement of kappa (23KDa) and lambda (45 KDa)free light chains levels, pre and post dialysis session, in patients undergoing high-flux dialysis versus HDF.

SECONDARY OUTCOMES:
Cumulative albumin loss | 1 day of hemodialysis session
  Assessment of cumulative dialysate albumin loss by measuring albumin spent in dialysate -hourly- in patients undergoing high flux dialysis versus HDF

CONTACTS AND LOCATIONS:
Overall Officials: Reem Sultan, M.Sc, Principal Investigator — Faculty of Medicine, Ain Shams Univeristy.; Hesham ElSayed, PhD, Study Chair — Faculty of Medicine, Ain Shams Univeristy; Magdy ElSharkawy, PhD, Study Chair — Faculty of Medicine, Ain Shams Univeristy; Waleed AbdelMohsen, PhD, Study Director — Faculty of Medicine, Ain Shams Univeristy; Shaimaa Zaki, PhD, Study Director — Faculty of Medicine, Ain Shams Univeristy; Ahmed Emara, PhD, Study Director — Faculty of Medicine, Ain Shams Univeristy
Locations (1):
- Ain Shams University Hospitals, Cairo, Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bourguignon C, Chenine L, Bargnoux AS, Leray-Moragues H, Canaud B, Cristol JP, Morena M. Hemodiafiltration improves free light chain removal and normalizes kappa/lambda ratio in hemodialysis patients. J Nephrol. 2016 Apr;29(2):251-257. doi: 10.1007/s40620-015-0207-z. Epub 2015 May 29. PMID 26022721
- [Background] Donati G, Moretti MI, Baraldi O, Spazzoli A, Capelli I, Comai G, Marchetti A, Sarma M, Mancini R, La Manna G. Removal of free light chains in hemodialysis patients without multiple myeloma: a crossover comparison of three different dialyzers. BMC Nephrol. 2016 Nov 25;17(1):193. doi: 10.1186/s12882-016-0405-5. PMID 27884120
- [Background] Lamy T, Henri P, Lobbedez T, Comby E, Ryckelynck JP, Ficheux M. Comparison between on-line high-efficiency hemodiafiltration and conventional high-flux hemodialysis for polyclonal free light chain removal. Blood Purif. 2014;37(2):93-8. doi: 10.1159/000357968. Epub 2014 Mar 1. PMID 24603634
- [Background] Maduell F. Hemodiafiltration versus conventional hemodialysis: Should "conventional" be redefined? Semin Dial. 2018 Nov;31(6):625-632. doi: 10.1111/sdi.12715. Epub 2018 May 29. PMID 29813181
- [Background] Nagai K, Tsuchida K, Ishihara N, Minagawa N, Ichien G, Yamada S, Hirose D, Michiwaki H, Kanayama HO, Doi T, Minakuchi J. Implications of Albumin Leakage for Survival in Maintenance Hemodialysis Patients: A 7-year Observational Study. Ther Apher Dial. 2017 Aug;21(4):378-386. doi: 10.1111/1744-9987.12526. Epub 2017 Apr 27. PMID 28452109
- [Background] van Gelder MK, Abrahams AC, Joles JA, Kaysen GA, Gerritsen KGF. Albumin handling in different hemodialysis modalities. Nephrol Dial Transplant. 2018 Jun 1;33(6):906-913. doi: 10.1093/ndt/gfx191. PMID 29106652
- [Background] Wolley M, Jardine M, Hutchison CA. Exploring the Clinical Relevance of Providing Increased Removal of Large Middle Molecules. Clin J Am Soc Nephrol. 2018 May 7;13(5):805-814. doi: 10.2215/CJN.10110917. Epub 2018 Mar 5. PMID 29507008
- [Background] Wolley MJ, Hutchison CA. Large uremic toxins: an unsolved problem in end-stage kidney disease. Nephrol Dial Transplant. 2018 Oct 1;33(suppl_3):iii6-iii11. doi: 10.1093/ndt/gfy179. PMID 30281131